CLINICAL TRIAL: NCT02086331
Title: Evaluation of Musculoskeletal Microcirculation With Ultrasound
Acronym: EMMU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/LO/0943; 13HH0684 (Other: Imperial College London)
Record Dates: First submitted 2014-01-09; First posted 2014-03-13 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Standardised Claudication Treadmill Test
Keywords: treadmill test
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (Active Comparator): Healthy volunteers, deemed to have normal metabolic and cardiovascular biology by trial criteria
  Interventions: Procedure: Contrast enhanced ultrasound; Behavioral: Treadmill test
- PAD (Active Comparator): Symptomatic peripheral arterial disease
  Interventions: Procedure: Contrast enhanced ultrasound; Behavioral: Treadmill test
- DM (Active Comparator): Symptomatic diabetic peripheral neuropathy
  Interventions: Procedure: Contrast enhanced ultrasound; Behavioral: Treadmill test

INTERVENTIONS:
Procedure: Contrast enhanced ultrasound — Infusion of microbubbles to enhance blood vessels in the leg for ultrasound
Behavioral: Treadmill test — Exposes you to exercise in a controlled environment. We will see if we can detect this change with our new ultrasound protocol
Procedure: Contrast enhanced ultrasound

SUMMARY:
This study aims to validate the use of Dynamic Contrast-Enhanced Ultrasound in measuring the blood supply to the muscles of the leg, and how this changes with exercise and vascular pathology.

DETAILED DESCRIPTION:
We propose a model for the use of Dynamic Contrast-Enhanced Ultrasound (DCEU) to directly evaluate the microcirculation of the musculoskeletal system. We believe that this will be a valuable research tool into diseases of the microcirculation, and in the future may also offer a clinical benefit by quantifying and monitoring disease over time and after intervention. It may also allow targeting of therapies towards those patients most at risk of ulcers and peripheral neuropathy, and those that would get the maximum benefit from these therapies.

ELIGIBILITY:
Group 1 - Healthy subjects Inclusion

* 18+ years old

Exclusion

* Personal history of diabetes or peripheral arterial disease, current pregnancy, previous surgery to the lower limb, heart attack within 4 weeks, or unstable angina

Group 2 - Peripheral arterial disease subjects Inclusion

* 18+ years old, radiological evidence of peripheral arterial disease (arterial doppler or angiogram), ankle-brachial pressure index (ABPI) 0.5-0.8

Exclusion

* Personal history of diabetes, current pregnancy, previous amputation, heart attack within 4 weeks, or unstable angina

Group 3 - Diabetic subjects Inclusion

* 18+ years old, with a clinical diagnoses of diabetes (1, 2)

Exclusion

- ABPI<0.9, previous amputation, current pregnancy or breastfeeding, heart attack within 4 weeks, or unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof AH Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early after the proof of concept stage. We showed that our methodology worked in healthy subjects, then ran out of time thus no participants were enrolled in either the "Symptomatic peripheral arterial disease" or "Symptomatic diabetic peripheral neuropathy" arms.
Groups:
- Healthy: Healthy participants
Period: Overall Study
Arm/Group | Healthy
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Poor recruitment. Trial closed early after 5 healthy recruits completed protocol.
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 23 [21 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Threshold of High to Low Frequency Ratio (Threshold HLFR)
Description: Please see published article for in depth method. This ratio is used to classify a given signal as either microbubble or noise. For a pixel containing a micro vessel, as microbubbles occasionally pass this otherwise dark pixel, its temporal signal is expected to have a higher proportion of lower frequency components than white noise. Consequently, the HLFR of the pixel is expected to be smaller than that of noise. A histogram of normalised HLFR shows two expected peaks (one noise, one bubbles). A threshold (Threshold HLFR) is determined to then separate the two peaks. this is done using a double Gaussian model, and where they intercept is deemed the Threshold HLFR.
Time Frame: Baseline, 20 minutes
Population: 5 recruits imaged and analysed. One recruit of five was excluded due to acquisition error
Measure: Number; unit: Threshold ratio (no units)
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4
Number analyzed (Participants) | 1 | 1 | 1 | 1
Threshold ratio (no units)
  At rest | 0.12 | 0.093 | 0.16 | 0.4
  After treadmill protocol, 20mins | 0.167 | 0.14 | 0.15 | 0.35
Statistical Analysis 1: Comparison: Subject 1 vs Subject 2 vs Subject 3 vs Subject 4; Test type: Other; Intraclass correlation of repeated measures - 0.96, p=0.08

2. Post Hoc Outcome: Average Percentage Change in Microbubble Track Density Measure (MTD)
Description: The number of pixels identified as having bubble signals was normalised by dividing by area of region of interest (ROI).
  MTD = pixels with microbubbles / area of ROI Used as a surrogate for active vascular density. The percentage change between rest and exercise (20 minute treadmill protocol) was calculated on each day
Time Frame: Test repeated on consecutive day to measure repeatability
Population: One subject out of five excluded for acquisition error
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Day 1 | Day 2
Number analyzed (Participants) | 4 | 4
% change from baseline | 138.2 (79.8) | 119.4 (62.7)

ADVERSE EVENTS:
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4 | Subject 5
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes